CLINICAL TRIAL: NCT02336958
Title: Ultrasound Guided Intermediate Cervical Plexus Block -Randomized Evaluation Concerning the Significance of Additional Perivascular Local Anesthetic Infiltration
Brief Title: Ultrasound Guided Intermediate Cervical Plexus Block and Additional Perivascular Local Anesthetic Infiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Research Center (Other)
Responsible Party: Principal Investigator, Dr.med.Ronald Seidel, MD, Helios Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A 2013-0075
Record Dates: First submitted 2015-01-02; First posted 2015-01-13 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Carotid Stenosis
Keywords: cervical plexus; regional anesthesia; ultrasound; carotid surgery
MeSH Terms: conditions — Carotid Stenosis | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaine (Active Comparator): Ultrasound guided intermediate cervical plexus block: 20ml ropivacaine 0.75%. Ultrasound guided perivascular/pericarotidal infiltration: 5ml ropivacaine 0.75%.
  Interventions: Drug: intermediate cervical plexus block ropivacaine; Drug: pericarotidal infiltration (active comparator) ropivacaine; Drug: jugular infiltration prilocaine
- saline (Placebo Comparator): Ultrasound guided intermediate cervical plexus block: 20ml ropivacaine 0.75%. Ultrasound guided perivascular/pericarotidal infiltration: 5ml saline 0.9%.
  Interventions: Drug: intermediate cervical plexus block ropivacaine; Drug: jugular infiltration prilocaine; Drug: pericarotidal infiltration (placebo comparator) saline

INTERVENTIONS:
Drug: intermediate cervical plexus block ropivacaine — 20ml ultrasound guided intermediate cervical plexus block.
Drug: pericarotidal infiltration (active comparator) ropivacaine — 5ml ropivacaine 0.75% (active comparator): pericarotidal infiltration.
  Arms: ropivacaine
Drug: jugular infiltration prilocaine — 5ml prilocaine 1% jugular infiltration for wound drainage.
Drug: pericarotidal infiltration (placebo comparator) saline — 5ml saline 0.9% (placebo comparator): pericarotidal infiltration.
  Arms: saline

SUMMARY:
For ultrasound guided intermediate cervical plexus block this randomized comparison is testing the hypothesis, that an additional perivascular infiltration is associated with increased block quality.

DETAILED DESCRIPTION:
The innervation of the neck is complex and involves the cervical and the brachial plexus as well as cranial nerves. So is the wall of the carotid arteries innervated by vagal and glossopharyngeal nerve as well as the sympathetic trunk. When carotid surgery was performed under regional anesthesia, so additional infiltration of local anesthetic by the surgeon was common, particularly during preparation of the carotid arteries.

Introduction of ultrasound guidance made it possible to guide the needle directly to the vascular wall. But this procedure is considered very demanding, because of guiding the needle in an anatomical region with artifacts (because of calcification), sudden movements (e.g. because of swallowing) and compromised coagulation (antithrombotic medication). On the other side there are no clinical data proving the benefit of an additional perivascular infiltration with local anesthetic. Therefore, this investigation is testing the hypothesis, that an additional perivascular infiltration is associated with increased block quality.

ELIGIBILITY:
Inclusion Criteria:

* carotid surgery (symptomatic and asymptomatic carotid stenosis)
* adult patients (18 years or older)
* ASA-risk-groups I-IV
* informed consent

Exclusion Criteria:

* drug allergy: local anesthetics
* pregnancy, lactation period
* participation in other studies
* addiction to drugs or alcohol
* non-cooperative patients
* no approval to regional anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Seidel, Dr.med., Principal Investigator — Helios Kliniken Schwerin, Klinik für Anästhesiologie und Intensivtherapie, Wismarsche Strasse 393-7, 19049 Schwerin, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine | Saline
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine | Saline | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (9.0) | 72.2 (7.7) | 71.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Required Supplementation of Local Anesthetic by Surgeon
Time Frame: during the intraoperative period
Measure: Number; unit: participants
Arm/Group | Ropivacaine | Saline
Number analyzed (Participants) | 20 | 20
participants | 13 | 13
Statistical Analysis 1: Comparison: Ropivacaine vs Saline; Test type: Superiority or Other; p = 1.0, Fisher Exact

2. Primary Outcome: Amount (ml) of Local Anesthetic Supplemented by Surgeon
Time Frame: during the intraoperative period
Measure: Mean (95% Confidence Interval); unit: ml
Arm/Group | Ropivacaine | Saline
Number analyzed (Participants) | 20 | 20
ml | 4.9 [2.2 to 7.6] | 3.7 [1.7 to 5.7]
Statistical Analysis 1: Comparison: Ropivacaine vs Saline; Test type: Superiority or Other; p = 0.459, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: during the intraoperative period
Arm/Group | Ropivacaine | Saline
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 17/20 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivacaine (N=20) | Saline (N=20)
definitive stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivacaine (N=20) | Saline (N=20)
temporarily hoarseness (Nervous system disorders) | 13 (13) | 11 (11)
temporarily dysphagia (Nervous system disorders) | 10 (10) | 5 (5)
cough (Nervous system disorders) | 11 (11) | 1 (1)
Horner syndrome (Nervous system disorders) | 8 (8) | 4 (4)
temporarily paresis of the hypoglossal nerve (Nervous system disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes